CLINICAL TRIAL: NCT05634577
Title: A Phase II Study to Evaluate the Efficacy and Safety of Pembrolizumab in Combination With Mitotane in Patients With Advanced Adrenocortical Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0705; NCI-2022-10009 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Adrenocortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Mitotane; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lead-in Phase (Experimental): Participants will first have a Lead-in Phase in which participants receive only mitotane. This will be 4 weeks long in most participants. Participants will then begin receiving pembrolizumab.
  Interventions: Drug: Mitotane; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Mitotane — Given by PO
Drug: Pembrolizumab — Given by vein (IV)

SUMMARY:
To learn if adding pembrolizumab to mitotane can help to control ACC. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Primary Objective(s), Hypothesis(es), and Endpoint(s):

(1) Objective: Assess the clinical efficacy of the combined use of MT with PEM in patients with advanced ACC.

Hypothesis: We hypothesize that adding PEM will enhance the clinical efficacy of MT. This additive/synergistic effect could be related to the intrinsic adrenolytic activity of MT that could lead to antigens exposures to immune cells. Furthermore, the cortisol lowering effect of mitotane is expected to alter the tumor microenvironment leading to a change the milieu of the tumor infiltrating immune cells to make ACC more susceptible to PEM. Also, cortisol lowering can reduce lymphocytes inhibition and enhances the efficacy of PEM.

Primary Endpoint: Overall response rate (ORR) assessed objectively using RECIST 1.1 criteria defined as the percentage of patients who have a partial or complete response to the combined treatment of MT plus PEM

Secondary Objective(s), Hypothesis(es), and Endpoint(s):

(1) Objective: Evaluate the safety and efficacy of the combined use of MT plus PEM in patients with advanced ACC.

Hypothesis: The optimal MT plasma levels have not been established prospectively in metastatic ACC. We hypothesize that mitotane level of 14-20 mg/L is associated with oncological responses, but we also anticipate that the combined use of PEM MT could be associated with responses at lower levels of MT which might be associated with more favorable AE profile of MT.

Secondary Endpoints:

1. Overall survival (OS), defined as the time from combination therapy to death from any cause.
2. Progression Free Survival (PFS), defined as the time from the start of combination therapy phase to disease progression or death from any cause.
3. Explore the association between MT level and response to therapy
4. Safety assessment by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0

Exploratory Objective(s):

(1) Objective: Correlate safety and efficacy data with steroid profile, immune markers and MT levels.

1. Obtain optional tumor biopsy prior to, during, and after treatment with MT/PEM combination to study immune markers such as infiltrating tumor lymphocytes, and other immune markers during therapy.
2. Study the changes in circulating markers (MT level, immune cytokines, steroid profile) in blood samples obtained prior to, during, and after treatment with MT/PEM combination

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of ACC will be enrolled in this study.
2. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and an additional 180 days after the last dose of study treatment and refrain from donating sperm during this period.
3. Female participants: A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period plus 180 days after the last dose of study treatment.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 10 days prior to the first dose of MT therapy.
7. Have adequate organ function as defined in the following table (Table 4). Specimens must be collected within 10 days prior to the start of study intervention.
8. The study will accept therapy naïve patients with metastatic ACC, patients who failed one prior line of therapy not including immunotherapy, patients who started MT within 4 weeks for metastatic disease, and patients who developed metastases while on adjuvant mitotane therapy. Patients who failed platinum-based chemotherapy combined with MT may be eligible to join the study at the discretion of the PI if their treatment ended > 6 months before consenting for this study or if did not achieve therapeutic MT levels during prior treatment (MT level ≥ 14 mg/L).
9. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen in the 28 days immediately preceding initiation of study treatment
10. Criteria for known Hepatitis B and C positive subjects

Hepatitis B and C screening tests are not required unless:

* Known history of HBV or HCV infection
* As mandated by local health authority

10.1 Hepatitis B positive subjects

* Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
* Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

10.2 Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Table 4 Adequate Organ Function Laboratory Values System Laboratory Value

* Hematological
* Absolute neutrophil count (ANC) ≥1500/µL
* Platelets ≥100 000/µL
* Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
* Renal
* Creatinine OR Measured or calculated b creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR

  ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
* Hepatic
* Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
* AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases) Coagulation
* International normalized ratio (INR) OR prothrombin time (PT)
* Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase);
* AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase);
* GFR=glomerular filtration rate; ULN=upper limit of normal.

a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

b Creatinine clearance (CrCl) should be calculated per institutional standard.

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to pembrolizumab treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent at the time of screening) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. Higher dose of steroid may be permitted as replacement doses while on mitotane therapy to follow acceptable standards of care while on mitotane Known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
11. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV) infection
14. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:
    * Known history of HBV and HCV infection
    * As mandated by local health authority
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
18. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mouhammed Habra, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients consented and one withdrew consent prior to immunotherapy (the key study intervention)
Groups:
- Combination Pembrolizumab With Mitotane: Active intervention
Period: Overall Study
Arm/Group | Combination Pembrolizumab With Mitotane
Started | 3
Completed | 1
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Pembrolizumab With Mitotane
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Assessment of tumor reduction by RECIST1.1 criteria
Time Frame: From time of active itervention (Combination therapy)
Population: Data were not collected for any participant due to study termination prior to participants' assessment at the pre-specified time points.
Arm/Group | Combination Pembrolizumab With Mitotane
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Time Frame: Overall survival (OS), defined as the time from combination therapy to death from any cause.
Population: as for outcome 1
Arm/Group | Combination Pembrolizumab With Mitotane
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival
Time Frame: Progression Free Survival (PFS), defined as the time from the start of combination therapy phase to disease progression or death from any cause.
Population: as for outcome 1
Arm/Group | Combination Pembrolizumab With Mitotane
Number analyzed (Participants) | 0

4. Secondary Outcome: Side Effects and Relationship Between Response and Drug Level
Time Frame: Explore the association between MT level and response to therapy Safety assessment by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Population: as for outcome 1
Arm/Group | Combination Pembrolizumab With Mitotane
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 1 year and 3 months
Description: Three particpants assessed for Adverse events
Arm/Group | Combination Pembrolizumab With Mitotane
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Pembrolizumab With Mitotane (N=3)
Nausea (Gastrointestinal disorders) | 1
Fever (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT05634577/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT05634577/ICF_000.pdf